CLINICAL TRIAL: NCT00003979
Title: Phase I and Pharmacokinetics Study to Determine the Safety of CHS 828 in Patients With a Solid Tumor on a Single Oral Dose Repeated Every 3 Weeks
Brief Title: CHS 828 in Treating Patients With Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16985; EORTC-16985
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — N-(6-chlorophenoxyhexyl)-N''-cyano-N''-4-pyridylguanidine

INTERVENTIONS:
Drug: CHS 828

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of CHS 828 in treating patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of oral CHS 828 in patients with solid tumors.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Determine a safe dose of this regimen for phase II evaluation.
* Determine the pharmacokinetic profile of this regimen in these patients.
* Determine any antitumor activity in these patients.

OUTLINE: Patients receive oral CHS 828 every 3 weeks. Treatment continues for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of CHS 828 until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity.

Patients are followed for up to 4 weeks.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor not amenable to standard therapy
* No symptomatic brain or leptomeningeal involvement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* Other liver function tests no greater than 2 times upper limit of normal (unless related to liver metastases)

Renal:

* Creatinine no greater than 1.4 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active bacterial infection
* No other nonmalignant disease
* No alcoholism, drug addiction, or psychiatric disorders
* Able to take oral medication

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas)
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy (6 weeks since extensive radiotherapy)
* No concurrent radiotherapy (except palliative radiotherapy)

Surgery:

* Not specified

Other:

* No other concurrent investigational drugs
* No other concurrent antitumor drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-04

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cerny, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (28):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Kaiser Franz Josef Hospital, Vienna
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Ludwig Institute for Cancer Research, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Herlev Hospital - University Hospital of Copenhagen, Copenhagen, Denmark
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
- Netherlands (5):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - Erasmus Medical Center, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Switzerland (3):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital - St. Gallen, Sankt Gallen
- United Kingdom (4):
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - C.R.C. Beatson Laboratories, Glasgow, Scotland

REFERENCES:
- [Result] Ravaud A, Cerny T, Terret C, Wanders J, Bui BN, Hess D, Droz JP, Fumoleau P, Twelves C. Phase I study and pharmacokinetic of CHS-828, a guanidino-containing compound, administered orally as a single dose every 3 weeks in solid tumours: an ECSG/EORTC study. Eur J Cancer. 2005 Mar;41(5):702-7. doi: 10.1016/j.ejca.2004.12.023. PMID 15763645